CLINICAL TRIAL: NCT01138202
Title: A Pilot Study of the Pharmacokinetics and Safety of Lopinavir/Ritonavir 400/100mg Bid Versus Lopinavir/Ritonavir 600/150 mg BID Combined With Nucleoside Analogue Reverse Transcriptase Inhibitors in HIV/TB Co-infected Patients Receiving Rifampicin Containing Anti-tuberculosis Therapy
Brief Title: Pharmacokinetics (PK) and Safety of 2 Different Doses of Lopinavir/Ritonavir in in HIV/Tuberculosis (TB) Co-infected Patients Receiving Rifampicin Containing Anti-tuberculosis Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: HIV-NAT 104
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections; Tuberculosis
Keywords: pharmacokinetics; safety; efficacy; Lopinavir/ritonavir; HIV/TB; rifampicin containing anti-tuberculosis therapy; Pharmacokinetics and safety of Lopinavir/ritonavir with rifampicin containing anti-tuberculosis therapy
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): boosted LPV/r 400/100 mg BID + 2 NRTI
  Interventions: Drug: LPV/r
- 2 (Experimental): boosted LPV/r 600/150 mg BID + 2 NRTI
  Interventions: Drug: LPV/r

INTERVENTIONS:
Drug: LPV/r — LPV/r 400/100 mg BID + 2 NRTI for arm 1 (total 48 weeks) LPV/r 600/150 mg BID + 2 NRTI for arm 2 (total 48 weeks)

SUMMARY:
To assess safety, efficacy and impact of Lopinavir/ritonavir 400/100mg bid or Lopinavir/ritonavir 600/150mg bid in combination with rifampicin-containing anti-TB therapy.

DETAILED DESCRIPTION:
Fixed dose combination of d4T+3TC+NVP (GPOvir) is widely used in Thai HIV infected since June 2002. The prevalence of NNRTI resistance has increased since 2005. Tuberculosis can develop following NNRTI-based regimen failure or after introduction of a new salvage regimen with a boosted PI (immune recovery syndrome). Although, Efavirenz based HAART is preferred in TB/HIV with rifampicin containing antituberculosis. However, Efavirenz could not be used in case of NNRTI failure, intolerance or toxicity. It remains unknown how to optimally treat HIV /TB in populations in which rifampicin has to be used. Moreover, Rifabutin which is recommended when use concomitant with boosted PI4, 5, is not feasible in Thailand and other developing countries due to cost, toxicity and dosing considerations. If ritonavir-boosted LPV demonstrates suitable pharmacokinetics, and is well tolerated, this regimen might prove extremely useful and could be widely implemented. LPV/r is potent and widely available boosted PI in National Health System in Thailand. We therefore believe that there is a strong rationale and impetus for the study of LPV/r 400/100 mg bid versus LPV/r 600/150 mg bid as a boosted-PI combination that in the presence of RMP, is able to produce a satisfactory PK profile associated with adequate antiretroviral potency, tolerability and efficacy .

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV positive after voluntary counseling and testing
2. Aged >18-60years of age
3. ARV naïve and NNRTI failure ( PI naive)
4. CD4+ cell count of <350 cells/mm3 at the time of diagnosed TB
5. ALT <5 times ULN
6. Serum creatinine <1.4 mg/dl
7. Hemoglobin >8 mg/L
8. TB is diagnosed and planned to receive stable doses of rifampicin-containing anti-TB therapy for at least a 2 week period after initiation of ART
9. No other active OI (CDC class C event), except oral candidiasis or disseminated MAC
10. Able to provide written informed consent

Exclusion Criteria:

1. Current use of steroid (except short course steroid for IRIS) and other immunosuppressive agents.
2. Current use of any prohibited medications related to drug pharmacokinetics.
3. Patients with current alcohol or illicit substance use that in the opinion of the site Principal Investigator would conflict with any aspect of the conduct of the trial.
4. Unlikely to be able to remain in follow-up for the protocol defined period.
5. Patients with proven or suspected acute hepatitis. Patients with chronic viral hepatitis are eligible provided ALT, AST < 5 x ULN.
6. Karnofsky performance score <30%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
plasma concentration level | 12 hours
  Percentage of plasma concentration level above an acceptable lower limit (lopinavir Cmin > 1 mg/L) at steady-state.

SECONDARY OUTCOMES:
identify toxicities | 48 weeks
  Toxicity of combined treatment for TB and HIV infections - the established DAIDS/ACTG toxicity grading scale of clinical and laboratory toxicities will be used.
CD4 | 48 weeks
  CD4 response (mean CD4 rise from baseline)
HIV RNA | 48 weeks
  HIV RNA response (% < 50 copies/ml at week 12, 24 and 48)
genotypic resistant | 48 weeks
  The emergence of NRTI and/or lopinavir genotypic resistant and its clinically

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- HIV-NAT Thai Red Cross AIDS Research Center, Bangkok, Thailand

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org